CLINICAL TRIAL: NCT05198648
Title: Trigeminal Nerve Cardiac Reflex During Resection of Cerebellopontine Angle Tumors and Postoperative Myocardial Injury: a Prospective Cohort Study
Brief Title: Trigeminal Nerve Cardiac Reflex During Resection of Cerebellopontine Angle Tumors and Postoperative Myocardial Injury
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Deputy chief of Department of Anesthesiology, Beijing Tiantan Hospital
Other Study IDs: 2021-12-12
Record Dates: First submitted 2021-12-13; First posted 2022-01-20 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Myocardial Injury; Trigeminal Cardiac Reflex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative myocardial injury
  Interventions: Other: Trigeminal cardiac reflex
- Non postoperative myocardial injury
  Interventions: Other: Non-trigeminal cardiac reflex

INTERVENTIONS:
Other: Trigeminal cardiac reflex — Trigeminal cardiac reflex occurred during the cerebellopontine angle tumor surgery.
  Groups: Postoperative myocardial injury
Other: Non-trigeminal cardiac reflex — No trigeminal cardiac reflex occurred during the cerebellopontine angle tumor surgery.
  Groups: Non postoperative myocardial injury

SUMMARY:
Myocardial injury after noncardiac surgery is significantly related to postoperative 30-day mortality. Trigeminal cardiac reflex is one of the main causes of perioperative cardiac emergency. Therefore, the investigators' aim is to test the hypothesis that trigeminal cardiac reflex associates postoperative myocardial damage in participants undergoing skull base tumor surgery. The investigators will observe the association between trigeminal cardiac reflex and myocardial injury by measuring the concentration of plasma high sensitivity cardiac troponin (hs-cTnT) in participants after skull base tumor surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective skull base tumor surgery.
* Age ≥ 18 years old.
* ASA class I to III.
* All those who sign the informed consent form.

Exclusion Criteria:

* Patients with severe heart disease (including patients with preoperative heart rate < 50 beats / min, severe arrhythmias, such as premature beats, paroxysmal supraventricular tachycardia, atrial flutter or fibrillation, patients with myocardial ischemia < 6 months, heart failure, myocarditis, pericarditis or cardiomyopathy).
* Patients unable to complete preoperative cardiac assessment.
* Patients with chronic kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged more than 18 years old with American Society of Anesthesiology status I to III who will be scheduled to receive elective skull base tumor surgery under general anesthesia. Patients with trigeminal cardiac reflex during surgery will be included in the exposure group while patients without trigeminal cardiac reflex during surgery will be included in the non-exposure group.
Sampling Method: Non-Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative myocardial injury | Postoperative 1 day.
  the elevation of plasma high sensitivity cardiac troponin I (hs-cTnI) caused by myocardial ischemia or injury (exclude other causes such as sepsis, pulmonary embolism, atrial fibrillation, etc). The blood samples before and within 24 hours after operation will be collected and measured by Roche's fourth generation hs-cTnI. It is commonly defined as an elevation as any value above the 99th percentile upper reference limit for each specific troponin I assay

SECONDARY OUTCOMES:
The duration time of trigeminal cardiac reflex during skull base tumor surgery. | The whole skull base tumor surgery procedure.
  The duration time of trigeminal cardiac reflex during skull base tumor surgery.

CONTACTS AND LOCATIONS:
Overall Officials: florapym766@163.com Peng, MD,Ph.D, Principal Investigator — Beijing Tian Tan Hospital
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No